CLINICAL TRIAL: NCT04734535
Title: Prospective, Randomized, Controlled, Multicenter, Clinical Investigation Evaluating the Safety of HEMOBLAST™ Bellows in Spine Surgery
Brief Title: Evaluation of Safety of HEMOBLAST Bellows in Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilon Technologies Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETC-2020-001
Record Dates: First submitted 2021-01-20; First posted 2021-02-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Surgical Bleeding
Keywords: Elective, spine surgery, bleeding control, hemostasis
MeSH Terms: interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Controlled, Multicenter, Clinical Investigation
Who Masked: Outcomes Assessor
Masking Description: data blinding to Sponsor, Independent Data Monitoring Committee, FDA reviewer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- investigational (Experimental): HEMOBLAST™ Bellows
  Interventions: Device: HEMOBLAST™ Bellows
- control (Active Comparator): absorbable gelatin sponge with thrombin
  Interventions: Device: absorbable gelatin sponge with thrombin

INTERVENTIONS:
Device: HEMOBLAST™ Bellows — Intraoperative bleeding during epidural spine surgery will be treated with HEMOBLAST™ Bellows
  Arms: investigational
Device: absorbable gelatin sponge with thrombin — Intraoperative bleeding during epidural spine surgery will be treated with absorbable gelatin sponge with thrombin
  Arms: control

SUMMARY:
The purpose of this clinical investigation in open, elective, spine surgery is to collect data to support the removal of the neurosurgical exclusion from the currently approved indication for the use of HEMOBLAST™ Bellows. This study is primarily designed to assess safety of the device for use in spine surgery, although efficacy information will also be captured and reported.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing open, elective, spine surgery
* Subject or an authorized legal representative is willing and able to give prior written informed consent for investigation participation
* Subject is 22 years of age or older
* Subject does not have an active or suspected infection at the surgical site
* Subject in whom the Investigator is able to identify a Target Bleeding Site (TBS) for which any applicable conventional means for hemostasis are ineffective or impractical
* Subject has a TBS with a Surface Bleeding Severity Scale (SBSS) score of 1, 2, or 3

Exclusion Criteria:

* Subject is undergoing an emergency surgical procedure
* Subject is undergoing a laparoscopic surgery
* Subject is undergoing a cervical spine surgery
* Subject is pregnant, planning on becoming pregnant during the follow-up period, or actively breast-feeding
* Subject has a platelet count < 100,000 per microliter or International Normalized Ratio > 1.5 within 4 weeks of surgery
* Subject receiving intravenous heparin within 12 hours before surgery or oral Coumadin within 2 days before surgery
* Subject receiving antiplatelet medications within 5 days prior to surgery
* Subject receiving aspirin within 7 days prior to surgery
* Subject has an active or suspected infection at the surgical site
* Subject has had or has planned to receive any organ transplantation
* Subject has a known sensitivity or allergy to bovine and/or porcine substance(s) or any other component(s) of the hemostatic agent
* Subject has a known sensitivity or allergy to Gadolinium
* The subject has a contra-indication for MRI or gadolinium contrast agent according to clinical guidelines, local regulations or manufacturer's recommendations
* Subject suffers from claustrophobia or fear of MRI, or has any contraindication to MRI (e.g., metal implants, spinal cord stimulator, etc. not suited to MRI)
* Subject has American Society of Anesthesiologists classification of > 4
* Subject has a life expectancy of less than 3 months
* Subject has a documented severe congenital or acquired immunodeficiency
* Subject has religious or other objections to porcine, bovine, or human components
* Subject is currently participating or has participated in another clinical trial within the past 30 days and is receiving/has received an investigational drug, device, or biologic agent
* Per investigator opinion subject is unable to fully cooperate with the study protocol.
* The product will be placed in at the site where the dura is open
* The product will be placed in the intradural or cranial space

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Unanticipated Adverse Device Effect (UADE) | 3 months follow-up
  incidence of UADE, for subjects treated with HEMOBLAST™, as determined by the Independent Data Monitoring Committee (IDMC).

SECONDARY OUTCOMES:
Adverse events (AE) | 3 months follow-up
  the proportion of AEs for subjects treated with HEMOBLAST™ compared to subjects treated with G+T.

OTHER OUTCOMES:
Hemostasis within 6 minutes | immediately after procedure
  Proportion of subjects achieving hemostasis within 6 minutes for HEMOBLAST™ subjects compared to G+T subjects
Operative time | immediately after procedure
  Operative time for HEMOBLAST™ subjects compared to G+T subjects
Length of stay | From procedure to discharge, estimated average = 36 hours
  Duration of hospitalization for HEMOBLAST™ subjects compared to G+T subjects
Blood transfusions | From procedure to discharge, estimated average = 36 hours
  Number of units of blood transfused intraoperatively for HEMOBLAST™ subjects compared to G+T subjects

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Schwab, MD, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - University of Southern California, Los Angeles, California
  - Indiana Spine Group, Carmel, Indiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spectrum Medical Inc, Danville, Virginia

IPD SHARING:
Plan to Share IPD: No